CLINICAL TRIAL: NCT01760395
Title: Complications in Inguinal Hernia Surgery - a Nationwide Registry Study
Brief Title: Complications in Inguinal Hernia Surgery
Status: Completed | Type: Observational
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Other Study IDs: NKCH-surg-010
Record Dates: First submitted 2012-12-31; First posted 2013-01-04 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Inguinal hernia repair is the most common procedure in general surgery. Even with acceptable complication rates, thousands of patients worldwide suffer from inguinal hernia surgery complications every year. In Finland, the Finnish Patient Insurance Centre (FPIC) receives reports from surgical complications. In this study, the database of FPIC is used to compare the complication profiles of open and laparoscopic inguinal hernia surgery with mesh.

ELIGIBILITY:
Inclusion Criteria:

* surgery between 2002 and 2010
* complicated inguinal hernia surgery reported to FPIC

Exclusion Criteria:

* none

Ages: 16 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Finnish patients having had complicated inguinal hernia surgery 2002-2010.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2002-01; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
surgical complication | 2 years

REFERENCES:
- [Derived] Kouhia S, Vironen J, Hakala T, Paajanen H. Open Mesh Repair for Inguinal Hernia is Safer than Laparoscopic Repair or Open Non-mesh Repair: A Nationwide Registry Study of Complications. World J Surg. 2015 Aug;39(8):1878-84; discussion 1885-6. doi: 10.1007/s00268-015-3028-2. PMID 25762240